CLINICAL TRIAL: NCT06008665
Title: Effects of Action Observation Therapy With Otago Exercises on Balance and Quality of Life in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Collaborators: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01345
Record Dates: First submitted 2023-07-10; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Balance; Distorted

STUDY DESIGN:
Who Masked: Participant
Masking Description: One of my group is experimental and the other one is controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action observation therapy with Otago exercise (Experimental): * Participants' Instructions:
  * Watch a video on a 22-inch screen.
  * Screen positioned 1 meter away from them.
  * Comfortably seated in a chair with armrests.
  * No following along or movement allowed.
  * Video Features: Model in the video is 70 years old or older. Model similar to the participants.
  * Video Viewing: Duration: 17 minutes (1 minute per video). Supervised by the same investigator. Quiet environment during observation.
  * Physical Training Session: Supervised by a therapist.
  * Duration: 35 minutes (2 minutes max per session).
  * Based on content from the video.
  * Action Observation Training: Activities during the physical education workshops featured in the videos.
  Interventions: Other: Action Observation Therapy and Otago Exercises
- Otago exercise (Active Comparator): * Strength Training Component:Knee Flexor, Knee Extensor, Hip Adductors, Ankle Planter Flexors, Ankle Dorsi Flexors
  * Balance Training Component:
  * Activities include: Walking backwards, Walking in a figure of eight, Heel-toe walking, Standing on one leg, Walking on the heels, Walking on the toes, Heel-toe walking backwards, Standing up from a sitting position, Walking up stairs.
  * Training Frequency and Guidance: Exercises conducted three times a week,Guidance provided by a therapist.
  * Training Session Duration: Each session lasts for 35-40 minutes.
  * Warm-up and Cool-down:5-minute warm-up before each session and 5-minute cool-down after each session.
  Interventions: Other: Otago Exercises

INTERVENTIONS:
Other: Action Observation Therapy and Otago Exercises — Strength Training Component:Knee Flexor, Knee Extensor, Hip Adductors, Ankle Planter Flexors, Ankle Dorsi Flexors
  Balance Training Component:
  Activities include: Walking backwards, Walking in a figure of eight, Heel-toe walking, Standing on one leg, Walking on the heels, Walking on the toes, Heel-toe walking backwards, Standing up from a sitting position, Walking up stairs.
  Training Frequency and Guidance: Exercises conducted three times a week,Guidance provided by a therapist.
  Training Session Duration: Each session lasts for 35-40 minutes. Warm-up and Cool-down:5-minute warm-up before each session and 5-minute cool-down after each session.
  Arms: Action observation therapy with Otago exercise
Other: Otago Exercises — Strength Training Component:Knee Flexor, Knee Extensor, Hip Adductors, Ankle Planter Flexors, Ankle Dorsi Flexors
  Balance Training Component:
  Activities include: Walking backwards, Walking in a figure of eight, Heel-toe walking, Standing on one leg, Walking on the heels, Walking on the toes, Heel-toe walking backwards, Standing up from a sitting position, Walking up stairs.
  Arms: Otago exercise

SUMMARY:
This study is to determine to see the effect of action observation therapy with otago exercise on Balance and Quality Of Life.

DETAILED DESCRIPTION:
This study is designed to reduce the Fall and balance problems and increase the quality of life in older adults. Balance, which declines with aging, is a complex sensory-motor process in which the visual, vestibular, and musculoskeletal systems work cooperatively to produce postural stability and loss of balance control causes falls, resulting in severe injuries, such as fractures, causing longstanding pain, lower quality of life, disability, and even death.

Interventions include balance and postural control that can help older people to avoid falling, through tai chi methods, gait training, strengthening exercises, and balance training programs.

The Otago Exercise Program comprises muscle strength exercises, balance training, and walking. The Otago workout program is based on individual tolerance, consisting of strengthening, balance, walking, and aerobic activities, and can be done at home environment Action observation is a cognitive intervention training strategy that involves observing other people's performance in order to promote motor learning.

Participants were instructed to watch a video on a screen while comfortably seated in a chair with armrests. They were not allowed to follow along or engage in any movement while watching the video. After the watching video of each component of otago exercises the exercises performed by participant based on the content of the video.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Participant experience fall > one time in last 6 months.
* Participants having Berg Balance score between 20 to 40

Exclusion Criteria:

* ●Abnormalities in visual, auditory, or vestibular system
* Limb defects
* History of recent fractures
* Participants with Cardiovascular, Cerebrovascular disease or traumatic brain injury and Epilepsy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline to 12th week
  The Berg Balance Scale is a testing tool with high validity and reliability used to measure balance. A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56. Score 0-20(High Risk of Fall), 21-40(Moderate Risk of Fall) and 41-54(Low Rosk of Fall)
Time Up and Go test | Baseline to 12th week
  The Timed Up and Go test is to identify mobility and balance impairments in older adults. Score ≥12 seconds (Risk of Fall)
Functional Reach Test | Baseline to 12th week
  The Functional Reach Test is a single item test developed as a quick screen for balance problems in older adults. Score >6 inches (High Risk of Fall), 6-10 inches (Risk of Fall)

SECONDARY OUTCOMES:
Short Form 36 | Baseline to 12th week
  The SF 36 is use to measure the Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Waqar Awan Awan, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No